CLINICAL TRIAL: NCT00823537
Title: Power-Assisted Therapeutic Electrical Stimulation to Upper Extremities in Acute Stroke Patients. A Randomized Controlled Trial.
Brief Title: Power-Assisted Therapeutic Electrical Stimulation to Upper Extremities
Acronym: TES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujita Health University (Other)
Responsible Party: Hitoshi Kagaya, Associate Professor, Fujita Health University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TES-RCT
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: therapeutic electrical stimulation

SUMMARY:
Power-assisted therapeutic electrical stimulation (TES) or conventional TES to upper extremities in acute stroke patients were performed in a randomized controlled trial. The changes in finger and hand function will be evaluated. The hypothesis is that a power-assisted TES is more effective than a conventional TES.

ELIGIBILITY:
Inclusion Criteria:

* acute or subacute phase of stroke

Exclusion Criteria:

* chronic phase of stroke

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)